CLINICAL TRIAL: NCT00682578
Title: Randomized Clinical Trial of the Efficacy and Safety of Dihydroartimisinine+Papiraquine (Artekin) Compared With First Line Drugs for Treatment of Vivax and Uncomplicated Falciparum Malaria in Afghanistan
Brief Title: A Comparative Study of Artekin With Standard Malarial Treatment Regimes in Afghanistan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Wellcome Trust (Other); Ministry of public Health Afghanistan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BKMAL0701
Record Dates: First submitted 2008-05-14; First posted 2008-05-22 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Uncomplicated Falciparum Malaria; Vivax Malaria
Keywords: falciparum malaria; vivax malaria; dihydroartemisinin-piperaquine
MeSH Terms: conditions — Malaria, Vivax; Malaria, Falciparum | interventions — artenimol; piperaquine; Pyrimethamine; Chloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Artekin (Experimental): Dihydroartemisinin+ Paperaquine (DHA+PPQ, Artekin)
  Interventions: Drug: Dihydroartemisinin + Piperaquine (Artekin)
- Standard treatment (Active Comparator): The standard treatment for uncomplicated falciparum and vivax malaria are as follows:
  Uncomplicated falciparum: artesunate-sulphadoxin/pyrimethamine Vivax malaria: chloroquine
  Interventions: Drug: artesunate-sulphadoxin/pyrimethamine, chloroquine

INTERVENTIONS:
Drug: Dihydroartemisinin + Piperaquine (Artekin) — An adult dose consists of four doses of two tablets, given at 0, 8, 24 and 48 h. The approximate total adult dose is 6/48 mg/kg (DHA/PPQ). For children, a dose of 1.6/12.8 mg/kg is given at the same time intervals; this dosage will be obtained by dissolving the tablets in 5 ml of water.
  Other Names: Artekin
  Arms: Artekin
Drug: artesunate-sulphadoxin/pyrimethamine, chloroquine — The standard treatment will be in accordance with that in Afghanistan
  Arms: Standard treatment

SUMMARY:
Malaria is a major public health problem in many provinces of Afghanistan the failure rate of chloroquine (CQ) and amodiaquine (AQ) treated Plasmodium falciparum(Pf) malaria has risen to more than 60% overall and as high as 90% in Jalalabad. CQ remains fully effective against P vivax, and sulphadoxine-pyrimethamine (SP) remains effective against P falciparum (10-15% of cases fail to cure). The current malaria treatment protocol still continuing CQ for P.vivax and adopted Artmisinine based combination therapy (ACT) for treating (Pf) malaria, as most than 50% malaria has being diagnosed clinically, so due to this and other operational reasons the protocol needs to be simplified.

By comparing 56 day PCR corrected cure rate of DHA-PPQ with the standard treatment regimen as primary objective and comparing the safety, gametocytecidal effect and parasite clearance time as secondary objectives, our study titled: Randomized, Open Label, controlled, non-inferiority clinical trial for comparison of Efficacy & safety, will provide scientific evidence to lead the simplification and improvement of the standard malaria treatment regimen in Afghanistan; to adopt a policy of treating both vivax and falciparum malaria with the same drug regimen.

With a significance level (α) = 0.05 and a power=80%, the calculated sample size is 274 per study arm. Therefore about1100 patients (274 per study-arm: 548 patients with falciaprum malaria and 548 patients with vivax malaria) will be recruited in Malaria reference Centers (MRCs) of three malaria endemic provinces (Nangarhar in the east, Thakhar in the north-east and Faryab in the north-west of country) after signing written inform consent form, according the inclusion and exclusion criteria and will be treated as out patients by giving the randomized drug dose under observation of study team and followed-up daily for 3 days (as treatment course of either arm is once daily dose for three days) and after than weekly up to day 56. and the study is planed to conducted in 3 provinces of Afghanistan for approximately 2 years.

Patients will be assessed clinically as well necessary laboratory tests will be performed and all the bio-medical findings will be recorded in special patient case record form, the electronic form of which will be broth to Trop. Med of Mahidol University for final analysis. The patients will be receiving the reasonable transportation cost for follow-up visits as well as one bed-net at the end of enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Uncomplicated falciparum or vivax malaria or mixed species infection, as confirmed in a peripheral blood slide.
* No signs of severe malaria
* Age over three months.
* Non-pregnant, (test for β-HCG in women of child-bearing age).
* Weight ≥5 kg
* Willingness to participate and written informed consent provided by the patient or in case of children by attending guardians/parents.
* Not enrolled in any other investigational drug study in the previous month

Exclusion Criteria:

* Clinical or laboratory features suggesting severe malaria.
* Known cardiac, renal, hepatic or other severe disease, or requirement for hospital treatment
* Recurrent vomiting.
* Not eligible for follow-up.
* Lactating mother
* Hyperparasitemia of P. falciparum > 100,000/µL
* Treatment with Artesunate or Chloroquine in the past one month, Fansidar in the past one and the half months and Artekin in past 3 months.

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1086 (Actual)
Dates: Start 2007-07 (Actual); Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
PCR corrected adequate clinical and parasitological response (PCR corrected 'adequate clinical and parasitological response' or ACPR) | Day 56

SECONDARY OUTCOMES:
Crude or PCR uncorrected ACPR | Day 56
Early treatment failure (failure to clear parasitaemia) | 7 days
fever clearance times | Days
parasite clearance times with no recrudescence over the observation period | days
gametocyte clearance times | weeks
Haemoglobin levels on day 14 compared to admission | day 14
safety and tolerability (rate and severity of adverse events) | day 56

CONTACTS AND LOCATIONS:
Overall Officials: Ghulam R Awab, MD, Principal Investigator — Provincial Malaria Control Centers (MRC)
Locations (4):
- Afghanistan (4):
  - Provincial Malaria Control Centers (MRC), Faryab
  - Provincial Malaria Control Centers (MRC), Jalalabad
  - Provincial Malaria Control Centers (MRC), Maymana
  - Provincial Malaria Control Centers (MRC), Takhar

REFERENCES:
- [Derived] Awab GR, Imwong M, Pukrittayakamee S, Alim F, Hanpithakpong W, Tarning J, Dondorp AM, Day NP, White NJ, Woodrow CJ. Clinical trials of artesunate plus sulfadoxine-pyrimethamine for Plasmodium falciparum malaria in Afghanistan: maintained efficacy a decade after introduction. Malar J. 2016 Feb 25;15:121. doi: 10.1186/s12936-016-1167-z. PMID 26917051
- [Derived] Awab GR, Pukrittayakamee S, Imwong M, Dondorp AM, Woodrow CJ, Lee SJ, Day NP, Singhasivanon P, White NJ, Kaker F. Dihydroartemisinin-piperaquine versus chloroquine to treat vivax malaria in Afghanistan: an open randomized, non-inferiority, trial. Malar J. 2010 Apr 21;9:105. doi: 10.1186/1475-2875-9-105. PMID 20409302